CLINICAL TRIAL: NCT01577368
Title: Efficacy and Safety of Piperacillin-Tazobactam Continuous Infusion vs Intermittent Infusion for Complicated or Nosocomial Pseudomonas Aeruginosa Infection or Suspected Infection
Brief Title: Piperacillin-Tazobactam Continuous Versus Intermittent Infusion for Pseudomonas Aeruginosa
Acronym: PiperTazo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: Ministerio de Sanidad y Política social (Unknown); Hospitales Universitarios Virgen del Rocío (Other); Hospital Universitario Virgen Macarena (Other); Hospital Son Espases (Other); Hospital Son Llatzer (Other); Complejo Hospitalario de Especialidades Juan Ramón Jimenez (Other); University Hospital Virgen de las Nieves (Other); Hospital General de Cataluña (Unknown); Hospital Infanta Sofia (Other); Hospital Universitario Ntra. Sra. de La Candelaria (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PiperTazo; 2010-024606-34 (EudraCT Number)
Record Dates: First submitted 2011-05-16; First posted 2012-04-13 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Pseudomonas Aeruginosa Infection
Keywords: Pseudomonas; Piperacillin; Beta-lactams; Continuous infusion; Intermittent infusion; Pharmacokinetics
MeSH Terms: conditions — Pseudomonas Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Piperacillin continuous infusion (Experimental): Piperacillin-Tazobactam 2gr (Loading dose DAY 1) plus Piperacillin-Tazobactam continuous infusion 8gr every 24 hours
  Interventions: Drug: Piperacillin-Tazobactam continuous infusion
- Piperacillin intermittent infusion (Active Comparator): Piperacillin-Tazobactam 4gr intermittent infusion 4gr every 8 hours
  Interventions: Drug: Piperacillin-Tazobactam intermittent infusion

INTERVENTIONS:
Drug: Piperacillin-Tazobactam continuous infusion — Piperacillin-Tazobactam 2gr (Loading dose DAY 1) plus Piperacillin-Tazobactam continuous infusion 8gr every 24 hours (DAY 1-14)
  Arms: Piperacillin continuous infusion
Drug: Piperacillin-Tazobactam intermittent infusion — Piperacillin-Tazobactam intermittent infusion 4gr every 8 hours (DAY 1-14)
  Arms: Piperacillin intermittent infusion

SUMMARY:
The main objective is to verify that the administration of piperacillin / tazobactam administered by continuous infusion to treat complicated infections or with known or suspected nosocomial isolation of Pseudomonas aeruginosa is superior in efficacy to a 30% higher dose administered in conventional short infusion.

The secondary objectives were compared between the following variables:

* Microbiological response at 3 days of starting treatment
* Time to microbiological cure
* Clinical response at 3 days of starting treatment
* Time to achieve defervescence
* To examine the relationship between pharmacokinetic variables and parameters of efficacy and safety
* To test the hypothesis that continuous infusion maintains adequate plasma drug levels compared with levels achieved with intermittent administration.
* Cost-effectiveness analysis
* Occurrence of adverse effects

To this end, we designed a multicenter, randomized, controlled, double blind, comparing both forms of administration in patients with complicated or nosocomial infection with or without isolation of Pseudomonas aeruginosa.

Patients who are candidates for inclusion are classified according to APACHE II and to have or not isolation of Pseudomonas aeruginosa. Subsequently be randomized to receive piperacillin-tazobactam by continuous infusion or short. Primary endpoint was measured as the ultimate effectiveness of treatment and other variables such as high efficiency, safety, pharmacokinetic and pharmacoeconomic.

ELIGIBILITY:
Inclusion Criteria:

* Complicated or Nosocomial Pseudomonas Aeruginosa Infection or Suspected Infection
* > 18 years and > 40 kg
* Negative pregnancy test for women within fertile period
* Informed consent signature

Exclusion Criteria:

* Life expectancy < 72 hr
* Central Nervous System (CNS) infection
* Ventilator-associated pneumonia
* Severe Neutropenia (<500 cells/ml)
* Acinetobacter baumannii or extended spectrum beta lactamase (ESBL) suspected infection
* Cystic fibrosis
* Shock
* Creatinine clearance < 20 ml/min
* Dialysis or hemoperfusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2011-05; Primary Completion 2014-01 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with satisfactory clinical response (cure or improvement) at the end of Piperacillin-Tazobactam treatment | 14 days
  * Clinical cure: complete resolution of all signs and symptoms of infection
  * Clinical improvement: resolution or improvement of most signs and symptoms of infection

SECONDARY OUTCOMES:
Proportion of patients with clinical response (cure or improvement) at 3 days | 3 days
  * Clinical cure: complete resolution of all signs and symptoms of infection
  * Clinical improvement: resolution or improvement of most signs and symptoms of infection
Proportion of patients with microbiological response | 3 days
  - Microbiological response: bacteriological eradication of causative organisms
Time to defervescence | 14 days
  - Time to the abatement of fever
Time to clinical cure | 14 days
Mortality | 28 days
Proportion of patients with adverse effects | 14 days & 60 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Seville, Spain